CLINICAL TRIAL: NCT04408729
Title: "PrEP My Way": A Novel PrEP Delivery System to Meet the Needs of Young African Women
Brief Title: PrEP My Way: A Novel PrEP Delivery System to Meet the Needs of Young African Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kenya Medical Research Institute (Other); Emory University (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Director of Research, Center for Global Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH122362 (NIH)
Record Dates: First submitted 2020-05-12; First posted 2020-05-29 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: HIV/AIDS
Keywords: prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP My Way intervention (Experimental): PrEP My Way is an intervention that involves peer-delivery of a kit containing PrEP and other sexual health services. Participants will be offered PrEP if HIV-negative per a point-of-care test, pregnancy testing, vaginal swabs for gonorrhea and chlamydia testing, condoms, and/or self-injection medroxyprogesterone, as desired.
  Interventions: Other: PrEP My Way
- Control (No Intervention): These participants will continue to receive PrEP at the clinic.

INTERVENTIONS:
Other: PrEP My Way — Intervention components may be modified pending the input from Aim 1. As currently planned, the peer delivering the PrEP My Way kit will be trained to provide basic education and support use of the kit components. The peer will also have a smart phone to show an instructional video. Participants will communicate with peers via mobile phones (e.g., SMS, WhatsApp) to arrange for kit delivery at Months 1, 3, and 6 via unmarked vehicles at home or a preferred safe site during reasonable hours. Two-way mobile phone communication will also be used to convey test results and provide on-going support and empowerment. Follow-up with the clinic will occur at Month 6 and as needed (e.g., treatment for positive tests).
  This intervention aims to increase adherence/persistence on PrEP. We hypothesize that removing the structural barriers and stigma associated with going to the clinic, women may be more likely to continue on PrEP.
  Arms: PrEP My Way intervention

SUMMARY:
The investigators will first develop, tailor, and refine PrEP My Way for use with young women in Kisumu, Kenya (Aim 1). The design firm will use a client-centered, iterative approach, involving up to 15 individual interviews and two focus group discussions (with up to 5 women each) to optimally design the PrEP My Way kit (with instructional materials) and peer delivery system (including communication and kit delivery plans). The investigators will then test the intervention for feasibility, acceptability, and preliminary impact on PrEP adherence and program retention (Aim 2). The study team will randomize 100 Kenyan women to PrEP My Way versus standard of care (i.e., clinic-based delivery of PrEP and sexual health services) and follow them for 6 months. Feasibility will be assessed by receipt of the kit at 1, 3, and 6 months and ability to use its components per protocol. Acceptability will be determined through a mixed-methods interview at 6 months. Preliminary impact will be evaluated by dried blood spot tenofovir levels (adherence) and kit use/clinic attendance at 6 months (retention) as primary outcomes. Mediators and moderators of PrEP use (e.g., empowerment and mental health) will be explored through questionnaires at baseline and 6 months.

DETAILED DESCRIPTION:
1. Develop PrEP My Way. Using a client-centered approach, the study team will iteratively conduct individual interviews and focus group discussions with up to 25 Kenyan women (age 16-24) to optimally design PrEP My Way (the kit with instructional materials) and peer delivery system (including phone communication and kit delivery plans).
2. Assess PrEP My Way for feasibility, acceptability, and preliminary impact on PrEP adherence and program retention. The investigators will randomize 100 Kenyan women (age 16-24) to PrEP My Way versus standard of care (i.e., clinic-based delivery of PrEP and sexual health services) and follow them for 6 months. Feasibility will be assessed by receipt of the kit at 1, 3, and 6 months and ability to use its components per protocol. Acceptability will be determined through a mixed-methods interview. Preliminary impact will be evaluated by dried blood spot tenofovir levels (adherence) and kit use/clinic attendance at 6 months (retention). Potential influencing and mediating socio-behavioral factors will be explored with questionnaires at 0 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Young woman (age 16-24 years); we will enroll emancipated minors (e.g., those who have not yet attained the age of legal competency as defined by state law, but who are entitled to treatment as if they had by virtue of assuming adult responsibilities, such as self-support, marriage, or procreation) per Kenyan national guidelines [39]) or 16-17 year-olds with parental consent
* Reported sexual activity within the past 3 months
* Interest in taking PrEP (actual PrEP uptake is not a requirement for Aim 1)
* Residence in the Kisumu region
* Phone ownership
* Ability to understand KiSwahili, DhoLuo, and/or English

Exclusion Criteria:

* Inability to provide informed consent (e.g., intoxication, mental disability)

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

RESULTS

PARTICIPANT FLOW:
Groups:
- PrEP My Way Intervention: PrEP My Way is an intervention that involves peer-delivery of a kit containing PrEP and other sexual health services. Participants will be offered PrEP if HIV-negative per a point-of-care test, pregnancy testing, vaginal swabs for gonorrhea and chlamydia testing, condoms, and/or self-injection medroxyprogesterone, as desired.
  PrEP My Way: Intervention components may be modified pending the input from Aim 1. As currently planned, the peer delivering the PrEP My Way kit will be trained to provide basic education and support use of the kit components. The peer will also have a smart phone to show an instructional video. Participants will communicate with peers via mobile phones (e.g., SMS, WhatsApp) to arrange for kit delivery at Months 1, 3, and 6 via unmarked vehicles at home or a preferred safe site during reasonable hours. Two-way mobile phone communication will also be used to convey test results and provide on-going support and empowerment. Follow-up with the clinic will occur at Month 6 and as needed (e.g., treatment for positive tests).
  This intervention aims to increase adherence/persistence on PrEP. We hypothesize that removing the structural barriers and stigma associated with going to the clinic, women may be more likely to continue on PrEP.
Period: Overall Study
Arm/Group | PrEP My Way Intervention | Control
Started | 75 | 75
Completed | 71 | 71
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEP My Way Intervention | Control | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21.6 [20.7 to 23.1] | 22.6 [20.9 to 23.9] | 22.3 [20.8 to 23.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 75 | 75 | 150
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: PrEP Adherence
Description: PrEP adherence as measured by detectable tenofovir-diphosphate (TFV-DP) in dried blood spots
Time Frame: Six months
Population: TFV-DP detection at 6 months per dried blood spots
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 75 | 75
Participants | 12 | 4

2. Secondary Outcome: Self-reported PrEP Adherence in the Past 30 Days
Description: PrEP adherence as measured by questionnaires at kit delivery.
Time Frame: Months 1, 3, 6 (intervention arm)
Population: Intervention participants reporting PrEP use at each kit delivery. Up to 75 participants could have taken PrEP at each time point; the number of participants analyzed at each time point is a subset of the 75, because not all participants chose to receive kits.
Measure: Mean (Full Range); unit: percentage of doses taken
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 75 | 0
percentage of doses taken
  Month 1: number analyzed (Participants) | 67 | 0
  Month 1 | 92 [17 to 100] |
  Month 3: number analyzed (Participants) | 59 | 0
  Month 3 | 79 [0 to 100] |
  Month 6: number analyzed (Participants) | 51 | 0
  Month 6 | 68 [0 to 100] |

3. Secondary Outcome: Number of Participants With PrEP Persistence (Kit Delivery/Pharmacy Refill)
Description: PrEP use as measured by PrEP receipt in the kit (intervention) or pharmacy pick up (control) at 6 months
Time Frame: At 6 months
Population: Study participants
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 75 | 75
Participants | 50 | 11

4. Secondary Outcome: Rates of STI Testing
Description: Testing for gonorrhea and chlamydia
Time Frame: Months 1, 3, and 6
Population: Participants who had STI testing done
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 75 | 75
Participants
  Month 1 | 67 | 0
  Month 3 | 64 | 0
  Month 6 | 62 | 0

5. Secondary Outcome: Rates of Hormonal Contraception
Description: Receipt of oral contraceptive pills or injections of medroxyprogesterone at least once among participants not using long-acting contraception (i.e., contraceptive implants or intrauterine devices)
Time Frame: Months 1, 3, and 6
Population: participants not using long-acting contraception (i.e., contraceptive implants or intrauterine devices)
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 61 | 52
Participants | 50 | 6

6. Secondary Outcome: Prevention-effective Adherence at 6 Months
Description: Detectable TFV-DP among women with ongoing HIV prevention needs, defined as meeting one or more of the following criteria: 1) PrEP use (per self-report and/or detectable TFVp-DP), 2) >1 concurrent sexual partner, 3) condomless sex, and 4) indication of "some/a lot of concern about getting HIV)
Time Frame: Measured at 6 months
Population: Women with ongoing HIV prevention needs, defined as meeting one of the following criteria: 1) PrEP use (per self-report and/or detectable TFVp-DP), 2) >1 concurrent sexual partner, 3) condomless sex, and 4) indication of "some/a lot of concern about getting HIV)
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 67 | 56
Participants | 12 | 4

7. Other Pre Specified Outcome: Feasibility of Intervention Use
Description: The PrEP My Way intervention will be considered feasible if >70% (35/50) participants 1) receive a kit at Months 1, 3, and 6; and 2) have a readable HIV test, usable vaginal swab, and self-injection of medroxyprogesterone, if desired, per protocol at >66% (2/3) of visits. The outcome indicates the number of participants at each time point who received a kit and were able to 1) read their HIV test (if testing was desired), 2) provide a vaginal swab that could be assessed for gonorrhea/chlamydia (if testing was desired), and 3) inject medroxyprogesterone (if the product was desired).
Time Frame: Six months
Population: Intervention participants
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 75 | 0
Participants
  Month 1 | 70 |
  Month 3 | 66 |
  Month 6 | 62 |

8. Other Pre Specified Outcome: Acceptability of Intervention
Description: The PrEP My Way intervention will be considered acceptable if >70% (35/50) participants rate 70% (7/10) items on the Systems Usability Scale (SUS) as "very good" or higher. The scores on the SUS are normalized on a scale 0-100 (higher scores indicate higher usability).
Time Frame: Six months
Population: Intervention participants completing the SUS at Month 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrEP My Way Intervention | Control
Number analyzed (Participants) | 68 | 0
units on a scale | 76 [68 to 85] |

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored/assessed from July 2021 - September 2022 (from the first enrollment through study completion for a total of 14 months, averaging 6 months per participant).
Arm/Group | PrEP My Way Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT04408729/Prot_SAP_000.pdf